CLINICAL TRIAL: NCT02395341
Title: The Effects of Cancer Treatment on Ovarian Function: A Longitudinal Study by the Oncofertility Consortium
Brief Title: The Longitudinal Ovarian Reserve Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 806409
Record Dates: First submitted 2015-03-17; First posted 2015-03-23 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Effects of Chemotherapy
Keywords: reproductive hormones; cancer survivors; endocrine function; antral follicle counts; female infertility due to diminished ovarian reserve; perimenopause; premature menopause
MeSH Terms: conditions — Menopause, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Postmenarchal female cancer patients scheduled to undergo cancer therapy may enroll in this study to assess changes in existing and novel surrogate measures of fertility potential before, during and after chemotherapy. Measures of fertility potential to be tested include ultrasound imaging for antral follicle counts and ovarian volumes, endocrine evaluation, and assessment of oxidative stress.

DETAILED DESCRIPTION:
Eligible women are asked to complete a structured interview, questionnaires, a monthly menstrual diary, a brief physical examination, a blood test, and an abdominal or pelvic ultrasound at baseline and at 3 month intervals following start of chemotherapy through 6 months post end of treatment.

Within subject changes in continuous variables (hormones, urinary isoprostane levels, ovarian volume, AFC) will be compared using paired t-tests (nonparametric tests as appropriate). Non-Gaussian-distributed variables will be logarithmically transformed prior to analysis. In general, changes from baseline to every 3 month assessment will be compared individually as well as changes from baseline to post treatment. In addition, regression models for repeated measures will be used to describe the pattern of change in these outcomes over time. Additional models will be constructed to adjust for potential confounding variables including age, chemotherapy type, dose and duration of treatment, radiation treatment, gonadotropin releasing hormone agonist use, and hormone use. Finally, regression models will be used to evaluate the association between changes in urinary isoprostane levels over the study with changes in endocrine measures.

ELIGIBILITY:
Inclusion Criteria:

* Females with the diagnosis of cancer schedules to be treated with chemotherapy and or radiation therapy.
* Age between 15-45 years.
* Post-menarchal.
* Presence of a uterus and both ovaries.
* Ability and willingness to comply with study protocol.
* Have given written informed concent (or assent with parental consent in minors), prior to any study-related procedure, not part of normal medical care, with the understanding that consent may be withdrawn byt he patient at any time without prejudice to their future medical care.

Exclusion Criteria:

* Current pregnancy.
* Lactation within the previous 3 months.
* Any medical condition other than cancer, with in the judgment of the investigator is known to be associated with premature ovarian failure (such as Turner's Syndrome or Fragile X) or ovulatory dysfunction (such as thyroid disease, adrenal dysfunction, Cushing's syndrome, hyperprolactinemia, and polycystic ovarian syndrome).

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be referred for this study by their primary oncologists. Eligible reproductive-aged girls and women newly diagnosed with cancer or another condition requiring chemotherapeutic intervention will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2009-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in reproductive hormone measures, during and after chemotherapy. | 18-24 months: pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  20 mls blood will be obtained at stated timepoints for determining levels of Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2), Inhibin B, and Anti-mullerian Hormone (AMH). In menstruating girls and young women hormone measures will be obtained during the early follicular phase of the menstrual cycle (days 1-4). In women with irregular cycles the testing will be done spontaneously without regard for the bleeding pattern.

SECONDARY OUTCOMES:
Change from baseline in ovarian volume during and after chemotherapy. | 18-24 months: Pelvic ultrasound will be performed at Pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  Ovaries will be measured in three dimensions. Uterine size and endometrial thickness will also be performed. The transvaginal approach is preferred, but transabdominal ultrasound will be performed in girls who do not feel comfortable with the transvaginal procedure.
Change from baseline in antral follicle counts during and after chemotherapy. | 18-24 months: Pelvic ultrasound will be performed at Pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  Antral Follicle Counts by size (2-5 mm, 6-9 mm, and >9 mm in diameter) will be determined.
Change in urinary isoprostane levels from baseline to 6 months after end of chemotherapy | 18-24 months: 24 hour urine collection will be performed at Pre-chemotherapy baseline and at the final study visit.
  24 hour urine collection will be analyzed to assess urinary 8,12-iso-iPF2alpha-VI isoprostane levels.
Change from baseline in menstrual characteristics | 18-24 months: Pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  Subjects are asked to document menstrual bleeding in a diary, noting duration of each menstrual period in days, bleeding intensity (spotting, light, moderate, heavy, flooding, none), and intervals between periods.
Change from baseline in menopausal symptoms | 18-24 months: Pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  The validated "Menopausal Symptom List" (MSL) will be used at each study visit to assess the presence or absence of menopausal symptoms during the past month, the frequency and severity of each symptom. Symptoms captured include: hot flashes, vaginal dryness, concentration/memory problems, irritability, mood swings, feeling sad, feeling anxious, trouble sleeping, aches, joint pain, headaches.
Change from baseline in quality of life measures | 18-24 months: Pre-chemotherapy baseline and at 3 month intervals from start of chemotherapy through 6 months after end of chemotherapy.
  One of two well validated and widely used questionnaires will assess Quality of Life measures: For adolescents 20 years of age or younger, the Minneapolis-Manchester Quality of Life (MMQL) - Adolescent Form will be administered. This questionnaire assesses demographics, physical functioning, cognitive functioning, psychological functioning, body image, social functioning, outlook on life, and intimate relations in cancer survivors. The MMQL is a 46 item validated, standardized self-report instrument designed to assess health related quality of life in adolescent survivors of cancer.
  Subjects over 20 years of age will be asked to complete a self report quality of life questionnaire entitled Assessing Quality of Life in Adult Cancer Survivors (QLACS). This questionnaire has been proven to be valid and reliable for comparing quality of life in adult cancer survivors and non-cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Clarisa R Gracia, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Penn Reproductive Research Unit, 3701 Market Street, Suite 810, Philadelphia, Pennsylvania
  - Penn Medicine at Radnor, 250 King of Prussia Road, Radnor, Pennsylvania